CLINICAL TRIAL: NCT06500260
Title: Natural History Study of Infants and Children With CNKSR2-Associated Neurodevelopmental Disorders and Epilepsy
Brief Title: CNKSR2 Natural History Study
Acronym: CNKSR2
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 22-35959
Record Dates: First submitted 2024-03-01; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Developmental Dysphasia; Epileptic Encephalopathy, Childhood-Onset; X-Linked Intellectual Disability
Keywords: X-linked Intellectual Disability; ESES; CSWS; CNKSR2; Epilepsy; Language Disorder
MeSH Terms: conditions — X-Linked Intellectual Disability; Epilepsy; Language Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective natural history study is being conducted to define the electroclinical, neurodevelopmental, and behavioral characteristics of CNKSR2 epilepsy aphasia syndrome (EAS) and intellectual disability (ID) in children aged 6 to 21 years old with CNKSR2 mutations.

The data collected from this study will serve as an external control to eventual clinical trials examining precision medicine investigational therapeutics that aim to improve the seizure burden and neurodevelopmental outcomes in patients with CNKSR2 EAS/ID.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 and 21 years (inclusive) at time of consent.
2. Confirmed CNKSR2 mutation, as demonstrated by genetic testing and confirmed by the investigators.
3. Confirmed intellectual disability or developmental delays, as defined by the American Academy of Pediatrics (Moeschler, J, et al. 2014).

Exclusion Criteria:

1. Known pathogenic or clinically suspected mutation in a seizure-associated gene besides CNKSR2.
2. Confirmed mutation in a gene besides CNKSR2 that is known to increase the severity of the seizure phenotype.
3. Known central nervous system structural abnormality confirmed by imaging scan of the brain that is not consistent with the clinical phenotype of CNKSR2 EAS / ID.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with CNKSR2 pathogenic mutation and characteristic features of CNKSR2 neurodevelopmental disorder and/or epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in functional connectivity within the epileptiform network using resting-state functional magnetic resonance imaging (fMRI). | Baseline, Month 12, Month 24
  Functional connectivity is unitless.
Change from baseline in functional connectivity within the language network using resting-state functional magnetic resonance imaging (fMRI). | Baseline, Month 12, Month 24
  Functional connectivity is unitless.
Change from baseline in cortical evoked response to self-produced speech as measured by voxel-wise source reconstructed brain activation using magnetoencephalography (MEG). | Baseline, Month 12, Month 24
  Voxel-wise source reconstructed brain activation assesses localized brain function by mapping neural activity at the voxel level. It is a unitless measure.
Change from baseline in cortical evoked response to altered auditory feedback during self-produced speech as measured by voxel-wise source reconstructed brain activation using magnetoencephalography (MEG). | Baseline, Month 12, Month 24
  Voxel-wise source reconstructed brain activation assesses localized brain function by mapping neural activity at the voxel level. It is a unitless measure.
Change from baseline in resting state brain activity as measured by voxel-wise source reconstructed brain activation using magnetoencephalography (MEG). | Baseline, Month 12, Month 24
  Voxel-wise source reconstructed brain activation assesses localized brain function by mapping neural activity at the voxel level. It is a unitless measure.
Change from baseline in resting state background brain activity during sleep as measured by phase lag index using electroencephalography (EEG). | Baseline, Month 12, Month 24
  Phase lag index ranges between 0 and 1 and is unitless. A phase lag index of zero indicates either no coupling or coupling with a phase difference centered around 0 mod π.
Change from baseline in spike-wave index during sleep as measured by percentage using electroencephalography (EEG). | Baseline, Month 12, Month 24
  Spike-wave index is the sum of all spike and slow wave minutes multiplied by 100 and divided by the total non-rapid eye movement sleep minutes.
Change from baseline in neurodevelopmental status as measured by Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III) scaled scores. | Baseline, Month 12, Month 24
  Higher scores indicate a better outcome (minimum score: 1, maximum score: 19).
Change from baseline in neurodevelopmental status as measured by the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSID-III) standard scores. | Baseline, Month 12, Month 24
  Higher scores indicate a better outcome (minimum score: 45, maximum score: 155).
Change from baseline in neurodevelopmental status as measured by the Wechsler Preschool and Primary Scale of Intelligence, 4th Edition (WPPSI-IV) composite scores. | Baseline, Month 12, Month 24
  Higher scores indicate a better outcome (minimum score: 40, maximum score: 160).
Change from baseline in neurodevelopmental status as measured by the Wechsler Preschool and Primary Scale of Intelligence, 4th Edition (WPPSI-IV) scaled scores. | Baseline, Month 12, Month 24
  Higher scores indicate a better outcome (minimum score: 1, maximum score: 19).
Change from baseline in neurodevelopmental status as measured by the Wechsler Abbreviated Scale of Intelligence, 2nd Edition (WASI-II) composite scores. | Baseline, Month 12, Month 24
  Higher scores indicate a better outcome (minimum score: 40, maximum score: 160).
Change from baseline in neurodevelopmental status as measured by the Wechsler Abbreviated Scale of Intelligence, 2nd Edition (WASI-II) T-scores. | Baseline, Month 12, Month 24
  Higher scores indicate a better outcome (minimum score: 20, maximum score: 80).
Change from baseline in neurodevelopmental status as measured by Parent Report Form of Vineland Adaptive Behavior Scales, 3rd Edition (Vineland-3) Adaptive Behavior Composite score and Domain scores. | Baseline, Month 12, Month 24
  Higher scores indicate a better outcome (minimum score: 20, maximum score: 140).
Change from baseline in neurodevelopmental status as measured by Parent Report Form of Vineland Adaptive Behavior Scales, 3rd Edition (Vineland-3) V-Scale Scores. | Baseline, Month 12, Month 24
  Higher scores indicate a better outcome (minimum score: 1, maximum score: 24).
Change from baseline in performance on the Receptive One-Word Picture Vocabulary Test, 4th Edition standard scores. | Baseline, Month 12, Month 24
  Higher scores indicate a better outcome (minimum score: < 55, maximum score: > 165).
Change from baseline in performance on the Expressive One-Word Picture Vocabulary Test, 4th Edition standard scores. | Baseline, Month 12, Month 24
  Higher scores indicate a better outcome (minimum score: < 55, maximum score: > 165).
Change from baseline in ADHD Rating Scale, 4th Edition (ADHD-RS-IV) inattention subscale raw scores. | Baseline, Month 6, Month 12, Month 18, Month 24
  Lower scores indicate a better outcome (minimum score: 0, maximum score: 9).
Change in hyperactivity as measured by ADHD Rating Scale, 4th Edition (ADHD-RS-IV) hyperactivity subscale raw scores. | Baseline, Month 6, Month 12, Month 18, Month 24
  Lower scores indicate a better outcome (minimum score: 0, maximum score: 9).
Change in physical functioning as measured by Pediatric Quality of Life Inventory (PedsQL) scale scores. | Baseline, Month 6, Month 12, Month 18, Month 24
  Lower scores indicate a better outcome (minimum score: 0, maximum score: 100).
Change in emotional functioning as measured by Pediatric Quality of Life Inventory (PedsQL) scale scores. | Baseline, Month 6, Month 12, Month 18, Month 24
  Lower scores indicate a better outcome (minimum score: 0, maximum score: 100).
Change in social functioning as measured by Pediatric Quality of Life Inventory (PedsQL) scale scores. | Baseline, Month 6, Month 12, Month 18, Month 24
  Lower scores indicate a better outcome (minimum score: 0, maximum score: 100).
Change in school functioning as measured by Pediatric Quality of Life Inventory (PedsQL) scale scores. | Baseline, Month 6, Month 12, Month 18, Month 24
  Lower scores indicate a better outcome (minimum score: 0, maximum score: 100).

CONTACTS AND LOCATIONS:
Overall Officials: Alex Fay, MD, PhD, Principal Investigator — alexander.fay@ucsf.edu
Locations (1):
- University of California, San Francisco (UCSF), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No